CLINICAL TRIAL: NCT03493763
Title: Study on Recurrence Monitoring of Hepatocellular Carcinoma With 5-Hydroxymethylcytosine Based on hmC-Seal Technology
Brief Title: Study on Recurrence Monitoring of Hepatocellular Carcinoma With 5-Hydroxymethylcytosine Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 5hmc HCC monitoring
Record Dates: First submitted 2018-04-01; First posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Recurrence Monitoring; 5-Hydroxymethylcytosine; Liquid biopsy; Cell-free DNA
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma cell-free DNA (cfDNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- serum AFP negative HCC patients: 1. Patients who received liver resection within 3 months;
  2. Hepatocellular carcinoma confirmed pathologically;
  3. Serum alpha-fetoprotein level lower than 20ng/ml before hepatectomy.
  Interventions: Diagnostic Test: 5hmC profile in plasma cell-free DNA after liver resection

INTERVENTIONS:
Diagnostic Test: 5hmC profile in plasma cell-free DNA after liver resection — Peripheral blood is drawn every 3 months after liver resection for 5hmC test (Time frame: 2 years or until tumor recurrence).

SUMMARY:
In this study, investigators aim to find out how plasma 5hmC level changes in hepatocellular carcinoma patients after liver resection, and determine whether 5hmC can be used as a biomarker for HCC recurrence monitoring.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary liver cancer and the third leading cause of cancer-related death worldwide. Liver resection is a common treatment for HCC. However, even after successful surgical resection, most patients suffered from recurrence or progression of the tumor. Because clinical staging systems cannot precisely predict the outcome of patients with HCC, it's of great interest to search biomarkers for HCC. Among them, alpha-fetoprotein (AFP) is the most well-studied. However, the applicability of AFP for HCC after surgical resection of tumor is still uncertain.

The discovery of cell-free DNA (cfDNA) originating from different tissues in the circulating blood has revolutionary potential for the clinic. Liquid biopsy-based biomarkers and detection tools offer substantial advantages over existing diagnostic and prognostic methods, including being minimally invasive. They thus have a cost-efficient potential to promote higher patient compliance and clinical convenience to enable dynamic monitoring.

5-hydroxymethylcytosine (5hmC) is the intermediate of active demethylation from 5-methylcytosine. 5hmC not only marks active demethylation but also serves as a relatively stable DNA mark that plays distinct epigenetic roles. Recent genome-wide sequencing maps of 5hmC in various mammalian cells and tissues support its role as a marker for gene expression. Previous studies have established 5hmC-Seal technology for 5hmC profiling in cfDNA and showed that the differentially enriched 5hmC regions in cfDNA are excellent markers for solid tumors.

In this study, investigators aim to find out how plasma 5hmC profile changes in hepatocellular carcinoma patients after liver resection, and determine whether 5hmC can be used as a biomarker for HCC recurrence monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received liver resection within 3 months;
2. Hepatocellular carcinoma confirmed pathologically;
3. Serum alpha-fetoprotein level lower than 20ng/ml before hepatectomy.

Exclusion Criteria:

1. Patients with macroscopic tumor remnants;
2. Patients with other diseases which may affect the observation mentioned here;
3. Patients with medical history of other malignant tumors;
4. Pregnant or nursing women.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be selected from patients who have received liver resection in the Liver Surgery Department of Zhongshan hospital.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Time of hepatocellular carcinoma recurrence | 2 years
  Time from the day of liver resection to the day of clinical diagnosis of recurrence

SECONDARY OUTCOMES:
5hmC level in recurrence-related cfDNA after liver resection | 2 years or until tumor recurrence
  Peripheral blood is drawn every 3 months after liver resection. 5hmc level in cfDNA in particular recurrence-related genes is tested by cfDNA sequencing and calculated by feature counts.
Serum alpha-fetoprotein level after liver resection | 2 years or until tumor recurrence
Adverse effect of 5hmC blood test | 2 years
  Any adverse effect of the test is to be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD&PhD, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No